CLINICAL TRIAL: NCT01858532
Title: A Randomized, Multicountry, Multicenter, Double-Blind, Parallel, Placebo-Controlled Study of the Effects of Atrasentan on Renal Outcomes in Subjects With Type 2 Diabetes and Nephropathy. SONAR: Study Of Diabetic Nephropathy With Atrasentan
Brief Title: Study Of Diabetic Nephropathy With Atrasentan
Acronym: SONAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-352; 2012-005848-21 (EudraCT Number)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetes; Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases | interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atrasentan (Active Comparator): 0.75 mg atrasentan once daily by mouth for up to 52 months
  Interventions: Drug: Atrasentan
- Placebo (Placebo Comparator): Placebo once daily by mouth for up to 52 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atrasentan — Film-coated tablet
  Other Names: ABT-627
  Arms: Atrasentan
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
The study objective was to evaluate the effect of atrasentan compared with placebo on time to doubling of serum creatinine (DBSC) or the onset of end-stage renal disease (ESRD) in participants with type 2 diabetes and nephropathy who were treated with the maximum tolerated labeled daily dose (MTLDD) of a renin-angiotensin system (RAS) inhibitor. In addition, the study assessed the effects of atrasentan compared with placebo on cardiovascular (CV) morbidity and mortality, urine albumin excretion, changes in estimated glomerular filtration rate (eGFR), as well as the impact on quality of life in participants with type 2 diabetes and nephropathy.

DETAILED DESCRIPTION:
This was a Phase 3, prospective, randomized, double-blind, enriched-population, placebo controlled, multicenter study in adult participants with type 2 diabetes and nephropathy. Participants who met the inclusion criteria for initial study entry and none of the exclusion criteria were eligible to proceed to the Run-In Period to optimize RAS inhibitor and diuretic doses. Following the Run-In Period, eligible participants entered the 6-week Enrichment Period in which all received atrasentan to determine their urinary albumin to creatinine ratio (UACR) response and to assess tolerability of atrasentan. Responders and nonresponders were then randomly assigned to receive atrasentan or placebo in the Double-Blind Treatment Period. The study was performed in 5 to 6 periods in the following sequence: Pre-Screening Period (optional); Screening Period (Visits S1 and S2); Run-In Period (up to 12 weeks; Visits R1 to R6); Enrichment Period (6 weeks; Visits E1 to E5); Double-Blind Treatment Period (randomization to final treatment visit); and Follow-Up Period (Final Treatment to F1 visit [45 days post treatment] and other post-treatment visits). The study was prematurely discontinued because of a lower than expected event rate for the renal composite endpoint, which was adjudicated by a blinded independent events adjudication committee (EAC).

ELIGIBILITY:
Inclusion Criteria:

* Participant, or legal representative, had voluntarily signed and dated an Informed Consent Form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study had been explained and the participant had the opportunity to ask questions. The informed consent must have been signed before any study-specific procedures were performed.
* Participant had type 2 diabetes (including participants with latent autoimmune diabetes or insulin-treated participants without a history of diabetic ketoacidosis who also had a negative anti-glutamic acid decarboxylase test AND an elevated post-prandial serum C-peptide level) and had been treated with at least one anti-hyperglycemic medication and an angiotensin-converting enzyme inhibitor (ACEi) or Angiotensin II receptor blocker (ARB; RAS inhibitor) for at least 4 weeks prior to the Screening S2 visit.
* For entry into the Run-In Period the participant must have satisfied the following criteria based on the Screening laboratory values:

  * Estimated glomerular filtration rate (eGFR) 25 to 75 mL/min/1.73 m^2 [until the eGFR cap on participants (approximately 300) with a baseline of > 60 mL/min/1.73 m^2 was reached] and a urine albumin creatinine ratio (UACR) greater than or equal to 300 and less than 5,000 mg/g (greater than or equal to 34 mg/mmol and less than 565 mg/mmol);
  * Serum albumin greater than or equal to 2.5 g/dL (25 g/L);
  * Brain natriuretic peptide (BNP) less than or equal to 200 pg/mL (200 ng/L);
  * Systolic blood pressure (SBP) greater than or equal to 110 and less than or equal to 180 mmHg;
  * Serum potassium greater than or equal to 3.5 mEq/L (3.5 mmol/L) and less than or equal to 6.0 mEq/L (6.0 mmol/L);
  * Participants on a maximum tolerated labeled daily dose (MTLDD) of a RAS inhibitor for greater than or equal to 4 weeks and on a diuretic at the time of screening and who satisfied the above criteria may have proceeded to the last visit in the Run-In Period (R6);
  * Participants already on a MTLDD of a RAS inhibitor for greater than or equal to 4 weeks and not on a diuretic (unless medically contraindicated) at the time of Screening were to start with a diuretic and participate in Run-In for at least 2 weeks.
* For entry into the Enrichment Period the participant must have satisfied the following criteria based on the last visit of the Run-In Period:

  * RAS inhibitor at the MTLDD for the previous 4 weeks with no adjustments of the dose;
  * Participants that were on a MTLDD RAS inhibitor and not on a diuretic (unless medically contraindicated) at the time of Screening must have been in Run-In for at least 2 weeks.
* For entry into the Double-Blind Treatment Period, participants must have satisfied the following criteria based on the last visit of the Enrichment Period:

  * RAS inhibitor at the MTLDD for the previous 6 weeks during the Enrichment Period with no adjustments of the dose;
  * Diuretic at any dose unless medically contraindicated or clinically intolerable in the investigator's judgement (i.e., hypotension or hypokalemia);
  * Participants must not have had a weight change greater than or equal to 3 kg from the beginning of Enrichment to the end of the Enrichment Period and absolute serum BNP greater than or equal to 300 pg/mL (300 ng/L) at the last Enrichment visit;
  * Participants must not have had an increase in serum creatinine greater than 0.5 mg/dL and greater than 20% increase from the beginning of Enrichment to the end of the Enrichment Period.

Exclusion Criteria:

A participant was not eligible for entry into the Run-in Period if he/she met any of the following criteria:

* Participant had a history of severe peripheral edema or facial edema requiring diuretics unrelated to trauma or a history of myxedema in the prior 4 weeks to the initial Screening S1 visit.
* Participant had a history of pulmonary hypertension, pulmonary fibrosis or any lung diseases requiring oxygen therapy (e.g., chronic obstructive pulmonary disease, emphysema).
* Participant had a documented diagnosis of heart failure, previous hospitalization for heart failure or current or constellation of symptoms (dyspnea on exertion, pedal edema, orthopnea, paroxysmal nocturnal dyspnea) felt to be compatible with heart failure, that was not explained by other causes, and for which there was a change in medication or other management directed at heart failure.
* Participant had known non-diabetic kidney disease (other than kidney stones).
* Participant had elevated liver enzymes (serum alanine aminotransaminase [ALT] and/or serum aspartate aminotransaminase [AST]) > 3 × the upper limit of normal (ULN).
* Participant had hemoglobin < 9 g/dL (90 g/L).
* Participant had a sensitivity to loop diuretics.
* Participant had a history of an allergic reaction or significant sensitivity to atrasentan (or its excipients) or similar compounds.
* Participant had a history of chronic gastrointestinal disease, which, in the Investigator's opinion, may have caused significant GI malabsorption.
* Participant had a history of secondary hypertension (i.e., hemodynamically significant renal artery stenosis, primary aldosteronism or pheochromocytoma).
* Participant had significant comorbidities (e.g., advanced malignancy, advanced liver disease) with a life expectancy of less than 1 year.
* Participant had clinically significant cerebrovascular disease (CVD) or coronary artery disease (CAD) within 3 months prior to the Screening S1 visit, defined as one of the following:

  * Hospitalization for MI or unstable angina; or
  * New onset angina with positive functional study or coronary angiogram revealing stenosis; or
  * Coronary revascularization procedure; or
  * Transient Ischemic Attack or Stroke.
* Participant had received any investigational drug including atrasentan within 3 months prior to the Screening S1 visit.
* Participant received dialysis treatments or was expected to receive dialysis or renal transplant within 6 months of screening.
* Participant was currently receiving rosiglitazone, moxonidine, aldosterone blockers, aliskiren or a combination of ACEi and ARB.
* Participant was a premenopausal woman defined as (for study purposes) any female subject with a menses in the past 2 years. For women who were < 50 years old, serum FSH must have been greater than 35 IU/L. Women who were surgically sterile or had a history of hysterectomy may not have necessarily be postmenopausal, and must also have had an FSH > 35 IU/L.
* Participant was at high risk for QT/QTc prolongation such as a family history of Long QT Syndrome, defined as QTc prolongation exceeding 450 ms in men, or 460 ms in women.
* Participant had type 1 diabetes.
* Participant was considered to be clinically unstable regarding general, metabolic or cardiovascular health as determined by the Investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5107 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Smeijer JD, de Vries ST, Kohan DE, Hou FF, Heerspink HJL. Sex differences in response to the endothelin receptor antagonist atrasentan in individuals with type 2 diabetes and chronic kidney disease: a post hoc analysis of the SONAR trial. Diabetologia. 2025 Mar;68(3):516-525. doi: 10.1007/s00125-024-06326-x. Epub 2024 Dec 11. PMID 39661119
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Smeijer JD, Kohan DE, Rossing P, Correa-Rotter R, Liew A, Tang SCW, de Zeeuw D, Gansevoort RT, Ju W, Lambers Heerspink HJ. Insulin resistance, kidney outcomes and effects of the endothelin receptor antagonist atrasentan in patients with type 2 diabetes and chronic kidney disease. Cardiovasc Diabetol. 2023 Sep 16;22(1):251. doi: 10.1186/s12933-023-01964-8. PMID 37716952
- [Derived] Chan KW, Smeijer JD, Schechter M, Jongs N, Vart P, Kohan DE, Gansevoort RT, Liew A, Tang SCW, Wanner C, de Zeeuw D, Heerspink HJL. Post hoc analysis of the SONAR trial indicates that the endothelin receptor antagonist atrasentan is associated with less pain in patients with type 2 diabetes and chronic kidney disease. Kidney Int. 2023 Dec;104(6):1219-1226. doi: 10.1016/j.kint.2023.08.014. Epub 2023 Aug 31. PMID 37657768
- [Derived] Smeijer JD, Koomen J, Kohan DE, McMurray JJV, Bakris GL, Correa-Rotter R, Hou FF, Januzzi JL, Kitzman DW, Kolansky DM, Makino H, Perkovic V, Tobe S, Parving HH, de Zeeuw D, Heerspink HJL. Increase in BNP in Response to Endothelin-Receptor Antagonist Atrasentan Is Associated With Incident Heart Failure. JACC Heart Fail. 2022 Jul;10(7):498-507. doi: 10.1016/j.jchf.2022.03.004. Epub 2022 May 4. PMID 35772861
- [Derived] Waijer SW, Gansevoort RT, Bakris GL, Correa-Rotter R, Hou FF, Kohan DE, Kitzman DW, Makino H, McMurray JJV, Perkovic V, Tobe S, Parving HH, de Zeeuw D, Heerspink HJL. The Effect of Atrasentan on Kidney and Heart Failure Outcomes by Baseline Albuminuria and Kidney Function: A Post Hoc Analysis of the SONAR Randomized Trial. Clin J Am Soc Nephrol. 2021 Dec;16(12):1824-1832. doi: 10.2215/CJN.07340521. Epub 2021 Dec 1. PMID 34853062
- [Derived] Koomen JV, Stevens J, Bakris G, Correa-Rotter R, Hou FF, Kitzman DW, Kohan DE, Makino H, McMurray JJV, Parving HH, Perkovic V, Tobe SW, de Zeeuw D, Heerspink HJL. Individual Atrasentan Exposure is Associated With Long-term Kidney and Heart Failure Outcomes in Patients With Type 2 Diabetes and Chronic Kidney Disease. Clin Pharmacol Ther. 2021 Jun;109(6):1631-1638. doi: 10.1002/cpt.2143. Epub 2021 Jan 5. PMID 33338269
- [Derived] Heerspink HJL, Parving HH, Andress DL, Bakris G, Correa-Rotter R, Hou FF, Kitzman DW, Kohan D, Makino H, McMurray JJV, Melnick JZ, Miller MG, Pergola PE, Perkovic V, Tobe S, Yi T, Wigderson M, de Zeeuw D; SONAR Committees and Investigators. Atrasentan and renal events in patients with type 2 diabetes and chronic kidney disease (SONAR): a double-blind, randomised, placebo-controlled trial. Lancet. 2019 May 11;393(10184):1937-1947. doi: 10.1016/S0140-6736(19)30772-X. Epub 2019 Apr 14. PMID 30995972

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5107 participants dosed in Enrichment Period (EP); 1441 prematurely discontinued Tx or did not proceed to Double-Blind Treatment Period per criteria. 3666 participants completed EP and proceeded to Double-Blind Treatment Period, along with 2 additional participants who discontinued study drug in EP but were randomized in error.
Groups:
- Intent-to-Treat (ITT) Responder Atrasentan: Participants who achieved at least 30% reduction in their albumin to creatinine ratio (UACR) in the Enrichment Period and were randomized to receive atrasentan in the Double-Blind Treatment Period
- Intent-to-Treat (ITT) Responder Placebo: Participants who achieved at least 30% reduction in their albumin to creatinine ratio (UACR) in the Enrichment Period and were randomized to receive placebo in the Double-Blind Treatment Period
- Intent-to-Treat (ITT) Non-responder Atrasentan: Participants who achieved < 30% reduction in their urinary albumin to creatinine ratio (UACR) in the Enrichment Period and were randomized to receive atrasentan in the Double-Blind Treatment Period
- Intent-to-Treat (ITT) Non-responder Placebo: Participants who achieved < 30% reduction in their urinary albumin to creatinine ratio (UACR) in the Enrichment Period and were randomized to receive placebo in the Double-Blind Treatment Period
Period: Overall Study
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo | Intent-to-Treat (ITT) Non-responder Atrasentan | Intent-to-Treat (ITT) Non-responder Placebo
Started | 1325 | 1323 | 509 | 511
Completed | 1144 | 1131 | 411 | 418
Not Completed | 181 | 192 | 98 | 93
Not completed — Adverse Event | 58 | 50 | 23 | 28
Not completed — Withdrew consent | 71 | 93 | 46 | 27
Not completed — Lost to Follow-up | 17 | 26 | 11 | 14
Not completed — Deterioration of medical status | 3 | 4 | 3 | 7
Not completed — Investigator request | 3 | 4 | 2 | 6
Not completed — Other, not specified | 29 | 15 | 13 | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Responders (participants who achieved at least 30% reduction in their albumin to creatinine ratio [UACR] in the Enrichment Period [EP]) and ITT Non-responders (Participants who achieved < 30% reduction in their UACR in the EP)
Groups:
- Total: Total of all reporting groups
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo | Intent-to-Treat (ITT) Non-responder Atrasentan | Intent-to-Treat (ITT) Non-responder Placebo | Total
Number analyzed (Participants) | 1325 | 1323 | 509 | 511 | 3668
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.64) | 64.7 (8.66) | 63.8 (9.12) | 63.6 (8.93) | 64.5 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331 | 352 | 127 | 136 | 946
  Male | 994 | 971 | 382 | 375 | 2722
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 30 | 29 | 7 | 10 | 76
  Asian | 446 | 455 | 143 | 154 | 1198
  Native Hawaiian or Other Pacific Islander | 9 | 9 | 7 | 3 | 28
  Black or African American | 73 | 76 | 36 | 39 | 224
  White | 753 | 744 | 313 | 300 | 2110
  More than one race | 14 | 10 | 3 | 5 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of a Component of the Composite Renal Endpoint in the Intent-to-Treat (ITT) Responder Set (as Randomized)
Description: Time to the first occurrence of a component of the composite renal endpoint was defined as doubling of serum creatinine (confirmed by a 30-day serum creatinine measurement) or the onset of end stage renal disease (estimated glomerular filtration rate [eGFR] less than 15 ml/min/1.73 m^2 confirmed by a 90-day eGFR measurement, receiving chronic dialysis, renal transplantation, or renal death). Only events adjudicated by the Events Adjudication Committee (EAC) were considered in defining this endpoint. Data are presented as number of participants with a primary renal composite event (first event per participant).
Time Frame: From randomization to individual end of observation, up to 53 months
Population: Intent-to-Treat (ITT) Responders (participants who achieved at least 30% reduction in their albumin to creatinine ratio [UACR] in the Enrichment Period [EP])
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo
Number analyzed (Participants) | 1325 | 1323
Participants | 79 | 105
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; The endpoint was analyzed using the stratified log-rank test for treatment comparison; Test type: Other; p = 0.029, Stratified log-rank test
Statistical Analysis 2: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; A Cox Proportional Hazards regression model with pre-specified covariates adjusted was used to estimate the hazard ratio of atrasentan to placebo and its 95% confidence interval; Test type: Other; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.654, 95% CI 2-sided [0.488 to 0.878]

2. Secondary Outcome: Time to a 50% Estimated Glomerular Filtration Rate Reduction in the Intent-to-Treat (ITT) Responder Set (as Randomized)
Description: The event of interest for this outcome was a 50% reduction in a participant's estimated glomerular filtration rate (eGFR) value as compared to baseline, confirmed by a repeated value at least 20 days apart. The event time was defined as the first time that a 50% reduction in eGFR was observed. Data are presented as number of participants with a 50% reduction in eGFR (first event per participant).
Time Frame: From randomization to individual end of observation, up to 53 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo
Number analyzed (Participants) | 1325 | 1323
Participants | 78 | 88
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; The endpoint was analyzed using the stratified log-rank test for treatment comparison; Test type: Other; p = 0.289, Stratified log-rank test
Statistical Analysis 2: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.112, Regression, Cox; Hazard Ratio (HR) = 0.779, 95% CI 2-sided [0.573 to 1.060]

3. Secondary Outcome: Time to Cardio-renal Composite Endpoint in the Intent-to-Treat (ITT) Responder Set (as Randomized)
Description: The composite event of interest for this outcome consisted of doubling of serum creatinine, end-stage renal disease (ESRD), cardiovascular (CV) death (including CV death and presumed CV death), nonfatal myocardial infarction (MI; heart attack) and nonfatal stroke. Presumed sudden cardiac death was included as a subcategory of presumed CV death. Only events adjudicated by the Events Adjudication Committee (EAC) were considered in defining this endpoint. Data are presented as number of participants with a cardio-renal composite event (first event per participant).
Time Frame: From randomization to individual end of observation, up to 53 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo
Number analyzed (Participants) | 1325 | 1323
Participants | 147 | 172
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; The endpoint was analyzed using the stratified log-rank test for treatment comparison; Test type: Other; p = 0.089, Stratified log-rank test
Statistical Analysis 2: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.049, Regression, Cox; Hazard Ratio (HR) = 0.801, 95% CI 2-sided [0.642 to 0.999]

4. Secondary Outcome: Time to First Occurrence of a Component of Composite Renal Endpoint for All Randomized Participants (Pooled)
Description: Time to the first occurrence of a component of the composite renal endpoint was defined as doubling of serum creatinine (confirmed by a 30-day serum creatinine measurement) or the onset of end stage renal disease (estimated glomerular filtration rate [eGFR] less than 15 ml/min/1.73 m^2 confirmed by a 90-day eGFR measurement, receiving chronic dialysis, renal transplantation, or renal death). Data for all randomized participants were pooled by treatment and analyzed. Data are presented as number of participants with a renal composite event (first event per participant).
Time Frame: From randomization to individual end of observation, up to 53 months
Population: Intent-to-treat population: participants who were randomized to receive either atrasentan or placebo during the Double-Blind Treatment Period
Measure: Count of Participants; unit: Participants
Groups:
- Intent-to-Treat (ITT) Atrasentan: All randomized participants who entered the Double-Blind Treatment Period and were randomized to receive atrasentan
- Intent-to-Treat Placebo: All randomized participants who entered the Double-Blind Treatment Period and were randomized to receive placebo
Arm/Group | Intent-to-Treat (ITT) Atrasentan | Intent-to-Treat Placebo
Number analyzed (Participants) | 1834 | 1834
Participants | 152 | 192
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) Atrasentan vs Intent-to-Treat Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.89]

5. Secondary Outcome: Time to the Cardiovascular Composite Endpoint in the Intent-to-Treat (ITT) Responder Set (as Randomized)
Description: The composite event of interest for this outcome was cardiovascular (CV) death (CV death, presumed CV death), nonfatal myocardial infarction (MI; heart attack), and nonfatal stroke. Presumed sudden cardiac death was included as a sub-category of presumed CV death. Only events adjudicated by the Events Adjudication Committee (EAC) were used. Data are presented as number of participants with a cardiovascular composite event (first event per participant).
Time Frame: From randomization to individual end of observation, up to 53 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intent-to-Treat (ITT) Responder Placebo: Intent-to-Treat (ITT) Responder Placebo: Participants who achieved at least 30% reduction in their albumin to creatinine ratio (UACR) in the Enrichment Period and were randomized to receive placebo in the Double-Blind Treatment Period
Arm/Group | Intent-to-Treat (ITT) Responder Atrasentan | Intent-to-Treat (ITT) Responder Placebo
Number analyzed (Participants) | 1325 | 1323
Participants | 72 | 81
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; The endpoint was analyzed using the stratified log-rank test for treatment comparison; Test type: Other; p = 0.446, Stratified log-rank test
Statistical Analysis 2: Comparison: Intent-to-Treat (ITT) Responder Atrasentan vs Intent-to-Treat (ITT) Responder Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.447, Regression, Cox; Hazard Ratio (HR) = 0.884, 95% CI 2-sided [0.643 to 1.215]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were reported from the time of study drug administration until 45 days after the last dose of study drug (up to 24 weeks for the All Atrasentan Set in the Enrichment Period; up to 54 months for the ITT sets in the Double-Blind Period)
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 45 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Enrichment Atrasentan: Participants who received at least one dose of atrasentan, including both Enrichment and Double-Blind Treatment Periods
- Double-Blind Atrasentan: All participants who received at least one dose of atrasentan during the Double-Blind Treatment Period
- Double-Blind Placebo: All participants who received at least one dose of placebo during the Double-Blind Treatment Period
Arm/Group | Enrichment Atrasentan | Double-Blind Atrasentan | Double-Blind Placebo
All-Cause Mortality (participants affected / at risk) | 25/5107 | 84/1829 | 79/1830
Serious Adverse Events (participants affected / at risk) | 292/5107 | 685/1829 | 626/1830
Other Adverse Events (participants affected / at risk) | 1781/5107 | 1043/1829 | 1038/1830
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrichment Atrasentan (N=5107) | Double-Blind Atrasentan (N=1829) | Double-Blind Placebo (N=1830)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7) | 27 (28) | 11 (15)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 5 (5) | 2 (2)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 3 (4)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 7 (7) | 34 (40) | 28 (29)
ADAMS-STOKES SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 4 (5) | 10 (11) | 10 (10)
ANGINA UNSTABLE (Cardiac disorders) | 4 (4) | 7 (7) | 3 (3)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 16 (17) | 10 (11)
ATRIAL FLUTTER (Cardiac disorders) | 2 (2) | 5 (5) | 2 (2)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 7 (7) | 2 (2)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
BRADYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 3 (3) | 4 (5) | 2 (2)
BUNDLE BRANCH BLOCK BILATERAL (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 3 (3) | 4 (4) | 5 (5)
CARDIAC FAILURE (Cardiac disorders) | 5 (5) | 19 (20) | 11 (11)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 4 (4) | 5 (6) | 4 (5)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 3 (3) | 5 (5) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 22 (22) | 37 (41) | 22 (23)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIORENAL SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 (6) | 29 (31) | 19 (20)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 3 (3) | 5 (5) | 2 (2)
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CYANOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERTENSIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 (3) | 4 (4) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 7 (7) | 13 (15) | 8 (8)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 9 (11) | 4 (4)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 4 (4) | 1 (1)
SINOATRIAL BLOCK (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
SINUS ARREST (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
GLUCOSE-6-PHOSPHATE DEHYDROGENASE DEFICIENCY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 7 (7)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERPARATHYROIDISM PRIMARY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
BLINDNESS TRANSIENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 3 (3) | 19 (19) | 10 (12)
CATARACT DIABETIC (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
CORNEAL EPITHELIUM DEFECT (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
CORNEAL OPACITY (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 2 (2) | 3 (4) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 3 (4) | 0 (0)
LAGOPHTHALMOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
PERIORBITAL OEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
RETINOPATHY PROLIFERATIVE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RHEGMATOGENOUS RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
TRACTIONAL RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VITREOUS ADHESIONS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 4 (4) | 9 (9) | 5 (7)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ANORECTAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETIC GASTROPATHY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
EROSIVE DUODENITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
GASTRIC DISORDER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
GASTRIC FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC MUCOSAL HYPERTROPHY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC POLYPS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 6 (6) | 3 (3)
GASTROINTESTINAL MUCOSAL DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 7 (7) | 2 (2)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
LYMPHOCYTIC OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1)
OBSTRUCTIVE PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
PANCREATIC DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (4)
PEPTIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
RECTAL POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
RECTAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ULCERATIVE GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3)
VOMITING (Gastrointestinal disorders) | 3 (3) | 7 (8) | 5 (5)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 2 (2)
BRAIN DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 7 (7) | 4 (4)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 3 (3) | 5 (5) | 4 (4)
DISEASE COMPLICATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
FEELING ABNORMAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
GENERALISED OEDEMA (General disorders) | 2 (2) | 3 (4) | 3 (3)
HYPOTHERMIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 3 (3) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 5 (5) | 3 (3)
NECROSIS (General disorders) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 4 (4) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 6 (6) | 3 (3)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 2 (2)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 1 (1) | 8 (8) | 5 (5)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0)
ULCER HAEMORRHAGE (General disorders) | 0 (0) | 0 (0) | 1 (1)
VASCULAR STENT STENOSIS (General disorders) | 1 (1) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (3)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 6 (6) | 3 (3)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 5 (5) | 3 (3)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
GALLBLADDER PERFORATION (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC LESION (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 6 (6) | 6 (7)
ABSCESS SOFT TISSUE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ACUTE SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
APPENDICITIS (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
ARTERIOSCLEROTIC GANGRENE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERIAL DIARRHOEA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
BILIARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BRAIN ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 9 (9) | 4 (4)
BRONCHITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 5 (5) | 14 (15) | 22 (24)
CELLULITIS GANGRENOUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CHRONIC TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DENGUE FEVER (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
DIABETIC FOOT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
DIABETIC GANGRENE (Infections and infestations) | 0 (0) | 2 (3) | 3 (3)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 4 (4) | 4 (4)
EMPHYSEMATOUS PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
ENDOPHTHALMITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTERITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
ERYSIPELAS (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 1 (3) | 4 (4) | 7 (7)
GAS GANGRENE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 8 (8) | 10 (10)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GRAFT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HELICOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTED SKIN ULCER (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTIVE EXACERBATION OF BRONCHIECTASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
JOINT ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LEPTOSPIROSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
MASTOIDITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
MEDICAL DEVICE SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MORGANELLA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NOSOCOMIAL INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 9 (11) | 10 (11)
OSTEOMYELITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PAROTID ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PERIODONTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PILONIDAL CYST (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 14 (14) | 54 (63) | 41 (43)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PROSTATIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PROSTATITIS ESCHERICHIA COLI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY TUBERCULOMA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 4 (4) | 16 (17) | 18 (18)
SEPSIS SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC EMBOLUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC NECROSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 5 (5) | 6 (6)
SIALOADENITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
TOXIC SHOCK SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (5) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 21 (21) | 12 (15)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
BLADDER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 7 (7) | 12 (12) | 5 (6)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
FOREIGN BODY IN GASTROINTESTINAL TRACT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (2)
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LISFRANC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SPINAL CORD INJURY CERVICAL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (3)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ULNAR NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WOUND NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLOOD BICARBONATE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 5 (5) | 7 (8)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM Q WAVE ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
HELICOBACTER TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
PROTEIN URINE PRESENT (Investigations) | 1 (1) | 1 (1) | 1 (1)
TROPONIN INCREASED (Investigations) | 0 (0) | 1 (1) | 2 (2)
URINE CYTOLOGY ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (7) | 11 (11) | 8 (8)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 3 (3) | 9 (9) | 7 (7)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
DIABETIC KETOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETIC METABOLIC DECOMPENSATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2 (2) | 9 (10) | 3 (3)
FLUID RETENTION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (3)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 8 (8) | 9 (11)
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5 (6) | 16 (18) | 16 (19)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 13 (13) | 22 (24) | 12 (14)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 6 (6)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (3)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
CHRONIC KIDNEY DISEASE-MINERAL AND BONE DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 4 (4)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISPLACEMENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 4 (4)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 3 (3)
MENISCAL DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 5 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8) | 16 (19)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SPINAL INSTABILITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPINAL LIGAMENT OSSIFICATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 1 (1)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
THORACIC SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ATYPICAL FIBROXANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 3 (3)
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
BLADDER CANCER STAGE I, WITH CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 3 (3)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
BRAIN NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CARCINOID TUMOUR PULMONARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 7 (7) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 2 (2)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GALLBLADDER CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4) | 6 (6)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)
HUERTHLE CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
INFLAMMATORY PSEUDOTUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LANGERHANS CELL SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT PALATE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTATIC CARCINOMA OF THE BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MUCINOUS ADENOCARCINOMA OF APPENDIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NEUROENDOCRINE TUMOUR OF THE LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
OESOPHAGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
OROPHARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OSTEOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 7 (7)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMYXOMA PERITONEI (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (4)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SINONASAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE HYPOPHARYNX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
TRANSITIONAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ACUTE MOTOR AXONAL NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
BRAIN STEM INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBELLAR HAEMATOMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 3 (3) | 8 (9)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
CEREBRAL THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5 (5) | 13 (14) | 14 (14)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETIC COMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETIC HYPERGLYCAEMIC COMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETIC HYPEROSMOLAR COMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOGLYCAEMIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 3 (3) | 2 (2) | 9 (10)
IVTH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MONONEUROPATHY MULTIPLEX (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCLONUS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
QUADRIPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 4 (6) | 2 (2)
SENILE DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 6 (6) | 11 (11)
THALAMIC INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 7 (7) | 7 (7)
VASCULAR DEMENTIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE CAPTURING ISSUE (Product Issues) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 1 (2) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DELUSIONAL DISORDER, SOMATIC TYPE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 19 (20) | 54 (56) | 36 (40)
AZOTAEMIA (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
BLADDER STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 9 (11) | 13 (13)
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 2 (2) | 17 (23) | 10 (11)
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 (0) | 19 (20) | 27 (30)
GLOMERULONEPHRITIS MEMBRANOUS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
HYDROURETER (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 4 (4) | 1 (1)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 5 (5) | 5 (5)
RENAL IMPAIRMENT (Renal and urinary disorders) | 3 (3) | 10 (11) | 13 (14)
RENAL VASCULITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 5 (7) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 7 (7)
EPIDIDYMAL CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 6 (6)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (11) | 9 (9)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) | 6 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
MEDIASTINAL CYST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 2 (2)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 4 (5)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 8 (8)
RESTRICTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
DIABETIC CHEIROARTHROPATHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (10) | 10 (10)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (10) | 3 (3)
OVERWORK (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
ANEURYSM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
ARTERIAL DISORDER (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIAL STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
ARTERITIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE INADEQUATELY CONTROLLED (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 4 (4) | 4 (4)
DIABETIC VASCULAR DISORDER (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DRY GANGRENE (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
EXTREMITY NECROSIS (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 9 (9) | 9 (9)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (2) | 1 (1) | 4 (4)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 4 (5) | 4 (5) | 4 (4)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 2 (2) | 7 (10)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 (2) | 2 (3) | 2 (2)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
VASCULAR OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrichment Atrasentan (N=5107) | Double-Blind Atrasentan (N=1829) | Double-Blind Placebo (N=1830)
ANAEMIA (Blood and lymphatic system disorders) | 180 (183) | 216 (241) | 127 (138)
DIARRHOEA (Gastrointestinal disorders) | 103 (108) | 99 (116) | 103 (110)
OEDEMA PERIPHERAL (General disorders) | 1148 (1273) | 534 (765) | 483 (666)
NASOPHARYNGITIS (Infections and infestations) | 145 (152) | 180 (274) | 169 (278)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 110 (114) | 106 (131) | 114 (140)
URINARY TRACT INFECTION (Infections and infestations) | 50 (51) | 93 (126) | 93 (135)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 77 (77) | 132 (159) | 143 (165)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 84 (85) | 101 (105) | 105 (106)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 126 (189) | 114 (193) | 120 (212)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 61 (62) | 88 (93) | 125 (133)
HYPERTENSION (Vascular disorders) | 78 (79) | 158 (179) | 218 (257)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT01858532/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT01858532/SAP_001.pdf